CLINICAL TRIAL: NCT00334828
Title: ACCESS: A Controlled Comparison of Eritoran Tetrasodium and Placebo in Patients With Severe Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E5564-G000-301; 2005-005537-35 (EudraCT Number)
Record Dates: First submitted 2006-06-06; First posted 2006-06-08 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Severe Sepsis
Keywords: Severe sepsis; septic shock; sepsis
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: eritoran tetrasodium
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: eritoran tetrasodium — Intravenous infusion at a total dose of 105 mg.
  Arms: 1
Drug: Placebo — Matching placebo; intravenous infusion.
  Arms: 2

SUMMARY:
The purpose of this study is to compare eritoran tetrasodium and placebo in patients with severe sepsis and to demonstrate a reduction of mortality from all causes.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age >= 18 years
* Confirmed early-onset severe sepsis, defined as:

  o---Objective evidence of infection likely to be caused by a bacterial or fungal pathogen

  o---Presence of at least 3 of 4 systemic inflammatory response syndrome (SIRS) criteria

  o---Sepsis-associated organ dysfunction
* Baseline Acute Physiology and Chronic Health Evaluation II (Apache II) Score of 21 to 37
* < 12 hours between onset of the first qualifying organ dysfunction and expected administration of study drug
* A commitment to full patient support

EXCLUSION CRITERIA:

* Pregnancy or breastfeeding
* Extensive (>20% Body Surface Area) third-degree burns
* Weight > 150 kg at admission
* Patients whose death from sepsis is considered imminent
* Patients not expected to survive for at least 2 months due to a pre-existing and uncorrectable medical condition, or those in a chronic vegetative state
* Patients with severe congestive heart failure
* Patients currently receiving immunosuppressive therapy such as cyclosporine, azathioprine, or cancer chemotherapy
* Patients with granulocyte counts < 1000/mm^3 unless the decreased count is believed to be due to sepsis
* Patients that required cardiopulmonary resuscitation in the 4 weeks prior to evaluation for enrollment
* Human immunodeficiency virus (HIV)-positive patients with CD4 count <= 50/mm^3 within 4 weeks of enrollment, or end-stage processes
* Patients with significant hepatic impairment, portal hypertension, or esophageal varices
* Patients who are expected to be treated with endotoxin-removal devices
* Patients with active cancer
* Patients receiving polymyxin B or colistin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2006-06; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
All-cause mortality at Day 28. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Dan Rossignol, Study Director — Eisai Inc.
Locations (251):
- United States (69):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Mesa, Arizona
  - Loma Linda, California
  - Marysville, California
  - Orange, California
  - San Diego, California
  - Santa Barbara, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Atlantis, Florida
  - Clearwater, Florida
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Oak Park, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Topeka, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Opelousas, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Pontiac, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Butte, Montana
  - Omaha, Nebraska
  - Englewood, New Jersey
  - Hackensack, New Jersey
  - Buffalo, New York
  - Mineola, New York
  - New Hyde Park, New York
  - New York, New York
  - Rochester, New York
  - Durham, North Carolina
  - Greenville, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Danville, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Columbia, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Roanoke, Virginia
  - Tacoma, Washington
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Santa Fe
- Australia (13):
  - New South Wales, New South Wales
  - St Leonards, New South Wales
  - Westmead, New South Wales
  - Queensland, Queensland
  - Southport, Queensland
  - Adelaide, South Australia
  - Woodville, South Australia
  - Heidelberg, Victoria
  - Melbourne, Victoria
  - Parkville, Victoria
  - Nedlands, Western Australia
  - Perth, Western Australia
  - Box Hill
- Austria (2):
  - Salzburg
  - Vienna
- Belgium (8):
  - Braine-l'Alleud
  - Brussels
  - Ghent
  - Liège
  - Mons
  - Ottignies
  - Seraing
  - Yvoir
- Brazil (7):
  - Belo Horizonte
  - Curitba
  - Fontaleza
  - Joinville
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Canada (12):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Windsor, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Québec, Quebec
- Chile (4):
  - Santiago
  - Temuco
  - Valdivia
  - Viña del Mar
- Czechia (5):
  - Brno
  - Havlíčkův Brod
  - Hradec Králové
  - Plyzen
  - Prague
- France (14):
  - Amiens
  - Besançon
  - Colombes
  - Corbeil-Essonnes
  - Evry Courcouronnes
  - La Roche-sur-Yon
  - La Tronche
  - Le Chesnay
  - Limoges
  - Montauban
  - Nîmes
  - Paris
  - Saint-Michel
  - Tours
- Germany (13):
  - Aachen
  - Berlin
  - Bonn
  - Cologne
  - Erfurt
  - Erlangen
  - Frankfurt
  - Geißen
  - Hanover
  - Jena
  - Krefeld
  - Ludwigshafen
  - München
- Hong Kong, Hong Kong
- Israel (10):
  - Afula
  - Hadera
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Petah Tikva
  - Tel Litwinsky
  - Ẕerifin
- Italy (9):
  - Bari
  - Busto Arsizio
  - Cesana Torinese
  - Milan
  - Monza
  - Novara
  - Pavia
  - Trieste
  - Verona
- Japan (30):
  - Aichi
  - Bunkyō City
  - Chūō
  - Fukuoka
  - Fukushima
  - Hachiōji
  - Hamamatsu
  - Hirosaki
  - Hiroshima
  - Iizuka
  - Kagoshima
  - Kamagaya
  - Kanagawa
  - Kishiwada
  - Kobe
  - Kochi
  - Kumamoto
  - Kyoto
  - Morioka
  - Osaka
  - Saga
  - Sapporo
  - Sendai
  - Shinagawa City
  - Suita
  - tabashi City
  - Ube
  - Utsunomiya
  - Yonago
  - Yotsukaidou
- Netherlands (10):
  - Amsterdam
  - Apeldoorn
  - Ede
  - Groningen
  - Leeuwarden
  - Rotterdam
  - s'Hertogenbosch
  - Tilburg
  - Utrecht
  - Zwolle
- Poland (6):
  - Bielsko-Biala
  - Groszisk Mazowiecki
  - Krakow
  - Lodz
  - Poznan
  - Warsaw
- Portugal (3):
  - Almada
  - Amadora
  - Lisbon
- South Africa (8):
  - Alberton
  - Cape Town
  - Centurion
  - Johannesburg
  - Kimberley
  - Parow
  - Pietermaritzburg
  - Roodepoort
- Seoul, South Korea
- Spain (9):
  - Alcala de Henares Madrid
  - Barcelona
  - Burgos
  - Cataluna
  - Getafe
  - Madrid
  - Sabadell
  - Santiago de Compostela
  - Tarragona
- Switzerland (3):
  - Bern
  - Geneva
  - Lausanne
- Taiwan (4):
  - Taichung
  - Taipei
  - Taoyuan District
  - Yung Kang City
- United Kingdom (7):
  - Birmingham
  - Leeds
  - Livingston
  - London
  - Nottingham
  - Plymouth
  - Southampton

REFERENCES:
- [Derived] Opal SM, Laterre PF, Francois B, LaRosa SP, Angus DC, Mira JP, Wittebole X, Dugernier T, Perrotin D, Tidswell M, Jauregui L, Krell K, Pachl J, Takahashi T, Peckelsen C, Cordasco E, Chang CS, Oeyen S, Aikawa N, Maruyama T, Schein R, Kalil AC, Van Nuffelen M, Lynn M, Rossignol DP, Gogate J, Roberts MB, Wheeler JL, Vincent JL; ACCESS Study Group. Effect of eritoran, an antagonist of MD2-TLR4, on mortality in patients with severe sepsis: the ACCESS randomized trial. JAMA. 2013 Mar 20;309(11):1154-62. doi: 10.1001/jama.2013.2194. PMID 23512062
- See also: Link to EUCTR results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2005-005537-35/results